CLINICAL TRIAL: NCT00052442
Title: A Phase II Study of 10-Propargyl-10-Deazaaminopterin (PDX) in Relapsed or Refractory Aggressive Non-Hodgkin's Lymphomas and Hodgkin's Disease
Brief Title: 10-Propargyl-10-Deazaaminopterin in Treating Patients With Recurrent or Refractory Non-Hodgkin's Lymphoma or Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000258425; MSKCC-02078; NCI-H02-0100
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Results first posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Lymphoma
Keywords: recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent mantle cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Mantle-Cell; Hodgkin Disease; Lymphoma, Follicular | interventions — 10-propargyl-10-deazaaminopterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 135 mg/m^2 Pralatrexate 1/2 weeks (Experimental): Pralatrexate (PDX) 135 mg/m^2 administered as an intravenous (IV) infusion over one hour into a side arm of a running intravenous infusion of normal saline for 1/2 weeks.
  Interventions: Drug: pralatrexate
- 30 mg/m^2 Pralatrexate 3/4 weeks (Experimental): PDX 30 mg/m^2 administered as an IV infusion over 15 minutes into a side arm of a running intravenous infusion of normal saline for 3/4 weeks.
  Interventions: Drug: pralatrexate
- 30 mg/m^2 Pralatrexate 6/7 weeks (Experimental): PDX 30 mg/m^2 administered as an IV infusion over 15 minutes into a side arm of a running intravenous infusion of normal saline for 6/7 weeks.
  Interventions: Drug: pralatrexate
- 45 mg/m^2 Pralatrexate 6/7 weeks (Experimental): PDX 45 mg/m^2 administered as an IV infusion over 15 minutes into a side arm of a running intravenous infusion of normal saline for 6/7 weeks.
  Interventions: Drug: pralatrexate
- 270 mg/m^2 Pralatrexate 2/4 weeks (Experimental): PDX (270 mg/m^2) administered as an IV bolus over 3-5 minutes into a side arm of a running intravenous infusion of normal saline for 2/4 weeks.
  Interventions: Drug: pralatrexate

INTERVENTIONS:
Drug: pralatrexate
  Other Names: Folotyn; 10-Propargyl-10-Deazaaminopterin (PDX)

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of 10-propargyl-10-deazaaminopterin in treating patients who have recurrent or refractory non-Hodgkin's lymphoma or Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of 10-propargyl-10-deazaaminopterin, in terms of objective response rate, duration of response, and time to disease progression, in patients with relapsed or refractory aggressive non-Hodgkin's lymphoma or Hodgkin's lymphoma.
* Determine the impact of pharmacokinetics on toxicity and drug elimination in patients treated with this drug.
* Determine the toxicity of this drug in these patients.
* Determine the effect of prior chemotherapy response duration on duration of response in patients treated with this drug.
* Correlate, if possible, the pharmacodynamics (area under the curve) of this drug with tumor response and toxicity (mucositis) in these patients.
* Correlate, if possible, intraerythrocytic folate or homocysteine levels with severity of mucositis in patients treated with this drug.
* Determine whether levels of the RFC-1 folate transporter, folylpolyglutamate synthetase, and folylpolyglutamate hydrolase are markers of response in patients treated with this drug.

OUTLINE: This is an open-label study.

Patients receive 10-propargyl-10-deazaaminopterin IV over 1 hour on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) may receive 2 additional courses beyond the CR.

PROJECTED ACCRUAL: A total of 39-72 patients (12-35 for cohort 1 and 17-37 for cohort 2) will be accrued for this study within 10-36 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Hodgkin's lymphoma or, using the World Health Organization (WHO) classification, aggressive non-Hodgkin's lymphoma including:

  * Large B- or T-cell lymphomas (including transformed lymphomas)
  * Mantle cell lymphoma
  * Immunoblastic lymphoma
* At least 1 unidimensionally measurable lesion

  * At least 2 centimeter (cm) by conventional techniques OR
  * At least 1 cm by spiral computerized tomography (CT) scan
  * Lymph nodes no greater than 1 cm in the short axis are considered normal
* Relapsed or refractory disease after first-line chemotherapy
* Cohort 1:

  * No more than 3 prior conventional cytotoxic chemotherapy regimens
  * Must have had at least a partial response (PR) lasting no more than 6 months or refractory disease
  * Patients with disease refractory to or relapsed less than 100 days from peripheral blood stem cell (PBSC) transplantation are not eligible
* Cohort 2:

  * No limit on prior treatment
  * Must have had at least a PR to the last therapy lasting at least 6 months
  * Patients who have received high-dose chemotherapy as part of peripheral blood stem cells (PBSC) transplantation are eligible if relapse occurred at least 100 days after transplantation
* No clinically significant pleural effusions or ascites
* No active brain or leptomeningeal metastases

  * Treated Central nervous system (CNS) disease allowed

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count greater than 1,000/mm^3
* Platelet count greater than 75,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* Aspartate aminotransferase/alanine aminotransferase (AST/ALT) no greater than 2.5 times ULN (4 times ULN if liver involvement)
* Alkaline phosphatase no greater than 5 times ULN

Renal

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 50 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No New York Heart Association class III or IV heart disease
* No unstable angina pectoris
* No cardiac arrhythmia
* No myocardial infarction, cerebrovascular accident, or transient ischemic attack within the past 6 months
* No history of orthostatic hypotension
* No ECG evidence of acute ischemia or significant conduction abnormality (e.g., bifascicular block or 2nd or 3rd degree atrioventricular blocks)
* No uncontrolled hypertension requiring active manipulation of antihypertensive medications
* No grade III or IV edema

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No ongoing or active infection

  * Febrile episodes up to 38.5° Celsius without signs of active infection allowed
* No other concurrent active cancer
* No other concurrent serious medical illness
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* At least 3 months since prior monoclonal antibody therapy (e.g., rituximab)

Chemotherapy

* See Disease Characterisitics
* At least 4 weeks since prior cytotoxic chemotherapy (6 weeks for mitomycin or nitrosoureas) and recovered

Endocrine therapy

* At least 7 days since prior steroids
* No concurrent steroids

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered

Surgery

* More than 4 weeks since prior major surgery

Other

* No prior antifolates
* No concurrent folic acid supplementation
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for human immunodeficiency virus (HIV)-positive patients
* No other concurrent investigational or commercial agents or therapies with the intent to treat the malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2002-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Owen A. O'Connor, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] O'Connor OA, Horwitz S, Hamlin P, Portlock C, Moskowitz CH, Sarasohn D, Neylon E, Mastrella J, Hamelers R, Macgregor-Cortelli B, Patterson M, Seshan VE, Sirotnak F, Fleisher M, Mould DR, Saunders M, Zelenetz AD. Phase II-I-II study of two different doses and schedules of pralatrexate, a high-affinity substrate for the reduced folate carrier, in patients with relapsed or refractory lymphoma reveals marked activity in T-cell malignancies. J Clin Oncol. 2009 Sep 10;27(26):4357-64. doi: 10.1200/JCO.2008.20.8470. Epub 2009 Aug 3. PMID 19652067

RESULTS

PARTICIPANT FLOW:
Groups:
- 135 mg/m^2 Pralatrexate 1/2 Weeks: Pralatrexate 135 mg/m^2 administered as an IV infusion over one hour into a side arm of a running intravenous infusion of normal saline for 1/2 weeks.
- 30 mg/m^2 Pralatrexate 3/4 Weeks: Pralatrexate 30 mg/m^2 administered as an IV infusion over 15 minutes into a side arm of a running intravenous infusion of normal saline for 3/4 weeks.
- 30 mg/m^2 Pralatrexate 6/7 Weeks: Pralatrexate 30 mg/m^2 administered as an IV infusion over 15 minutes into a side arm of a running intravenous infusion of normal saline for 6/7 weeks.
- 45 mg/m^2 Pralatrexate 6/7 Weeks: Pralatrexate 45 mg/m^2 administered as an IV infusion over 15 minutes into a side arm of a running intravenous infusion of normal saline for 6/7 weeks.
- 270 mg/m^2 Pralatrexate 2/4 Weeks: Pralatrexate 270 mg/m^2 administered as an IV bolus over 3-5 minutes into a side arm of a running intravenous infusion of normal saline for 2/4 weeks.
Period: Overall Study
Arm/Group | 135 mg/m^2 Pralatrexate 1/2 Weeks | 30 mg/m^2 Pralatrexate 3/4 Weeks | 30 mg/m^2 Pralatrexate 6/7 Weeks | 45 mg/m^2 Pralatrexate 6/7 Weeks | 270 mg/m^2 Pralatrexate 2/4 Weeks
Started | 16 | 3 | 27 | 11 | 15
Completed | 16 | 3 | 27 | 11 | 15
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all patients with at least one dose of pralatrexate.
Groups:
- 135 mg/m2 Pralatrexate 1/2 Weeks: Pralatrexate 135 mg/m^2 administered as an IV infusion over one hour into a side arm of a running intravenous infusion of normal saline for 1/2 weeks.
- 30 mg/m2 Pralatrexate 3/4 Weeks: Pralatrexate 30 mg/m^2 administered as an IV infusion over 15 minutes into a side arm of a running intravenous infusion of normal saline for 3/4 weeks.
- 30 mg/m2 Pralatrexate 6/7 Weeks: Pralatrexate 30 mg/m^2 administered as an IV infusion over 15 minutes into a side arm of a running intravenous infusion of normal saline for 6/7 weeks.
- 45 mg/m2 Pralatrexate 6/7 Weeks: Pralatrexate 45 mg/m^2 administered as an IV infusion over 15 minutes into a side arm of a running intravenous infusion of normal saline for 6/7 weeks.
- 270 mg/m2 Pralatrexate 2/4 Weeks: Pralatrexate 270 mg/m^2 administered as an IV bolus over 3-5 minutes into a side arm of a running intravenous infusion of normal saline for 2/4 weeks.
- Total: Total of all reporting groups
Arm/Group | 135 mg/m2 Pralatrexate 1/2 Weeks | 30 mg/m2 Pralatrexate 3/4 Weeks | 30 mg/m2 Pralatrexate 6/7 Weeks | 45 mg/m2 Pralatrexate 6/7 Weeks | 270 mg/m2 Pralatrexate 2/4 Weeks | Total
Number analyzed (Participants) | 16 | 3 | 27 | 11 | 15 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (16.1) | 54.3 (14.4) | 55.7 (16.5) | 52.7 (11.4) | 57.1 (15.1) | 54.1 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 10 | 7 | 5 | 28
  Male | 12 | 1 | 17 | 4 | 10 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 2 | 2 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 3 | 2 | 3 | 11
  White | 10 | 0 | 21 | 5 | 9 | 45
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 1 | 2 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Per Response Evaluation Criteria in T-cell and B-cell Lymphoma for target lesions and assessed using computerized tomography (CT) and or Positron emission tomography CT (PET CT) by local investigators: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=50% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 135 mg/m^2 Pralatrexate 1/2 Weeks | 30 mg/m^2 Pralatrexate 3/4 Weeks | 30 mg/m^2 Pralatrexate 6/7 Weeks | 45 mg/m^2 Pralatrexate 6/7 Weeks | 270 mg/m^2 Pralatrexate 2/4 Weeks
Number analyzed (Participants) | 16 | 3 | 27 | 11 | 15
Participants | 15 | 3 | 27 | 11 | 15

2. Secondary Outcome: Toxicities of Pralatrexate
Description: Adverse events; number of patients with at least one adverse events reported.
Time Frame: 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 135 mg/m^2 Pralatrexate 1/2 Weeks | 30 mg/m^2 Pralatrexate 3/4 Weeks | 30 mg/m^2 Pralatrexate 6/7 Weeks | 45 mg/m^2 Pralatrexate 6/7 Weeks | 270 mg/m^2 Pralatrexate 2/4 Weeks
Number analyzed (Participants) | 16 | 3 | 27 | 11 | 15
Participants | 16 | 3 | 27 | 11 | 15

ADVERSE EVENTS:
Arm/Group | 135 mg/m^2 Pralatrexate 1/2 Weeks | 30 mg/m^2 Pralatrexate 3/4 Weeks | 30 mg/m^2 Pralatrexate 6/7 Weeks | 45 mg/m^2 Pralatrexate 6/7 Weeks | 270 mg/m^2 Pralatrexate 2/4 Weeks
Serious Adverse Events (participants affected / at risk) | 8/16 | 1/3 | 15/27 | 10/11 | 10/15
Other Adverse Events (participants affected / at risk) | 8/16 | 2/3 | 12/27 | 1/11 | 5/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 135 mg/m^2 Pralatrexate 1/2 Weeks (N=16) | 30 mg/m^2 Pralatrexate 3/4 Weeks (N=3) | 30 mg/m^2 Pralatrexate 6/7 Weeks (N=27) | 45 mg/m^2 Pralatrexate 6/7 Weeks (N=11) | 270 mg/m^2 Pralatrexate 2/4 Weeks (N=15)
Stomatitis (Gastrointestinal disorders) | 6 (6) | 0 (0) | 3 (3) | 3 (3) | 3 (3)
Vomitting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutropenia & Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 2 (2)
General Disorders (General disorders) | 0 (0) | 0 (0) | 6 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 135 mg/m^2 Pralatrexate 1/2 Weeks (N=16) | 30 mg/m^2 Pralatrexate 3/4 Weeks (N=3) | 30 mg/m^2 Pralatrexate 6/7 Weeks (N=27) | 45 mg/m^2 Pralatrexate 6/7 Weeks (N=11) | 270 mg/m^2 Pralatrexate 2/4 Weeks (N=15)
Nausea (Gastrointestinal disorders) | 8 (8) | 2 | 12 | 1 | 5

LIMITATIONS AND CAVEATS:
Study completed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No